CLINICAL TRIAL: NCT01979965
Title: Ranolazine Effects on Ischemic Mitral Regurgitation Severity in Patients With Cardiac Resynchronization Therapy
Brief Title: Effect of Ranolazine on Valvular Disease in Patients With Pacemakers
Acronym: REIN-MR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IN-US-259-0173
Record Dates: First submitted 2013-10-23; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Mitral Regurgitation
Keywords: Mitral Regurgitation; cardiac resynchronization therapy; ranolazine; maximal medical therapy; ischemic cardiomyopathy
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active drug (Active Comparator): Ranolazine therapy for three months
  Interventions: Drug: Ranolazine (Active drug)
- Sugar Pill (Placebo Comparator): sugar pill therapy for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine (Active drug) — Ranolazine therapy for three months
  Other Names: Ranexa
  Arms: Active drug
Drug: Placebo — Placebo therapy for three months
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to find out whether mitral regurgitation (or a leaky heart valve) caused by ischemic heart disease (decreased blood flow to heart muscle) will improve after administration of ranolazine.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cardiomyopathy AND
* Moderate or severe mitral regurgitation AND
* Cardiac resynchronization therapy (CRT) ≥ 3 months prior to enrollment AND
* Maximal Medical Therapy (ACE-Inhibitor, beta blocker, aldosterone antagonist, diuretic, aspirin, statin)

Exclusion Criteria:

* nonischemic cardiomyopathy
* active heart failure
* current ranolazine therapy
* congenital heart disease
* mechanical valve prostheses
* vegetation/endocarditis
* significant pulmonary disease
* peripheral vascular disease
* trivial or mild mitral regurgitation
* creatinine clearance < 30 mL/min
* liver cirrhosis
* strong inhibitors of CYP3A (including ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir)
* strong inducers of CYP3A (including rifampin, rifapentine, phenobarbital, phenytoin, carbamazepine and St.John's wort)
* Strong P-glycoprotein inhibitors (including cyclosporine, verapamil, and quinidine)
* Initial QTc interval ≥ 440msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
effective regurgitant orifice by echocardiography | Day T = 90 days
proximal isovelocity surface area by echocardiography | T = 90 days

SECONDARY OUTCOMES:
Seattle Angina Questionnaire | T = 0 days, and T = 90 days
Rose Dyspnea Scale | T = 0 days, and T= 90 days

OTHER OUTCOMES:
Adverse Reactions | T = 90 day

CONTACTS AND LOCATIONS:
Overall Officials: Raj Baljepally, MD, Principal Investigator — University Cardiology
Locations (1):
- University Cardiology, Knoxville, Tennessee, United States

REFERENCES:
- See also: University Cardiology — http://utcardiology.com